CLINICAL TRIAL: NCT06316388
Title: Anatomical and Functional Outcomes After Vitrectomy in Eyes With Tractional Diabetic Macular Edema
Brief Title: Outcomes After Vitrectomy in Eyes With Tractional Diabetic Macular Edema
Status: Not yet recruiting | Type: Observational
Sponsor: Rehab Azzam (Other)
Responsible Party: Sponsor-Investigator, Rehab Azzam, Principle investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: TDME
Record Dates: First submitted 2024-03-09; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: vitrectomy — pars plana vitrectomy

SUMMARY:
1. assessment the outcomes of vitrectomy on retinal function by mf-ERG (multifocal electroretinogram) and anatomy by OCT (optical coherence tomography) in patients with tractional diabetic macular edema (TDME) .
2. To correlate the postoperative corrected distance visual acuity (CDVA) with the mf-ERG and OCT findings following vitrectomy surgery for TDME.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is one of the leading causes of vision loss worldwide [1]. In 2010, DR affected more than 93 million individuals worldwide, 28 million of whom experienced vision-threatening DR[2].

Diabetic macular edema (DME) is a common cause of visual loss in diabetic retinopathy (DR) and is a complication in any stages of DR including proliferative diabetic retinopathy (PDR)[3].

The terms vitreous traction maculopathy, vitreous induced diabetic macular edema and maculopathy due to posterior hyaloid traction are synonymous and describe a pattern of diabetic maculopathy which is characterized by: (1) The absence of complete posterior vitreous detachment; (2) An increased retinal thickness in the center of the macula, and (3) a characteristic reflex of the vitreoretinal interface[4]. there are multiple factors in the vitreomacular interface including ERM, taut posterior cortices, vitreoschisis, PVD, and adhesions [5]. Anomalous PVD generates antero-posterior and tangential traction forces at the vitreo-retinal interface that act upon the inner and outer retinal layers [6]. Until recently, the only treatment option available for VMA was vitrectomy[7].

Few studies have used the multifocal electroretinogram (mfERG) technique to investigate the effects of vitrectomy on macular visual function for DME [8]. Mf-ERG is an objective electrophysiologic technique that measures the electrical changes in the central retinal area. This technique accurately assess the electrophysiologic activity in multiple retinal areas, and gives us a topographic charting of retinal function [9] .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years; type 1 or 2 diabetes
* TDME as the indication for vitrectomy; central foveal thickness (CFT) ≥300 µm as measured by spectral-domain optical coherence tomography (SD-OCT) , We defined VMIA on OCT as ERM, anomalous vitreomacular adhesions, or both , ), and possible visual acuity impairment attributed to foveal thickening due to DME.

Exclusion Criteria:

* A history of other retinal diseases; or active ocular inflammation or infection or glaucoma .
* Eyes with macular edema from etiologies other than diabetes
* Dense refractive media opacity before and after surgery, such as dense cataract, vitreous hemorrhage which can conceal fundus visualization and OCT measurements
* Central retinal ischemia detected by intravenous fluorescein angiograms.
* A history of vitrectomy
* A visual acuity worse than 1\60 and the duration of tractional ERM is more than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: eyes with tractional diabetic macular edema
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-03-11 (Estimated)

PRIMARY OUTCOMES:
assessment the outcomes of vitrectomy on retinal function in patients with tractional diabetic macular edema | baseline
  assessment the outcomes of vitrectomy on retinal function by mf-ERG (multifocal electroretinogram) in patients with tractional diabetic macular edema
assessment the outcomes of vitrectomy on retinal anatomy in patients with tractional diabetic macular edema | Baseline
  assessment the outcomes of vitrectomy on retinal anatomy by OCT (optical coherence tomography) in patients with tractional diabetic macular edema

SECONDARY OUTCOMES:
correlation CDVA with mf-ERG and OCT finding | baseline
  To correlate the postoperative corrected distance visual acuity (CDVA) with the mf-ERG and OCT findings following vitrectomy surgery for TDME.

CONTACTS AND LOCATIONS:
Overall Officials: ehab wasfi, prof, Study Chair — Assiut University

REFERENCES:
- [Background] Lee R, Wong TY, Sabanayagam C. Epidemiology of diabetic retinopathy, diabetic macular edema and related vision loss. Eye Vis (Lond). 2015 Sep 30;2:17. doi: 10.1186/s40662-015-0026-2. eCollection 2015. PMID 26605370
- [Background] Yau JW, Rogers SL, Kawasaki R, Lamoureux EL, Kowalski JW, Bek T, Chen SJ, Dekker JM, Fletcher A, Grauslund J, Haffner S, Hamman RF, Ikram MK, Kayama T, Klein BE, Klein R, Krishnaiah S, Mayurasakorn K, O'Hare JP, Orchard TJ, Porta M, Rema M, Roy MS, Sharma T, Shaw J, Taylor H, Tielsch JM, Varma R, Wang JJ, Wang N, West S, Xu L, Yasuda M, Zhang X, Mitchell P, Wong TY; Meta-Analysis for Eye Disease (META-EYE) Study Group. Global prevalence and major risk factors of diabetic retinopathy. Diabetes Care. 2012 Mar;35(3):556-64. doi: 10.2337/dc11-1909. Epub 2012 Feb 1. PMID 22301125
- [Background] Romero-Aroca P, Baget-Bernaldiz M, Pareja-Rios A, Lopez-Galvez M, Navarro-Gil R, Verges R. Diabetic Macular Edema Pathophysiology: Vasogenic versus Inflammatory. J Diabetes Res. 2016;2016:2156273. doi: 10.1155/2016/2156273. Epub 2016 Sep 28. PMID 27761468
- [Background] Lewis H, Abrams GW, Blumenkranz MS, Campo RV. Vitrectomy for diabetic macular traction and edema associated with posterior hyaloidal traction. Ophthalmology. 1992 May;99(5):753-9. doi: 10.1016/s0161-6420(92)31901-3. PMID 1594222
- [Background] Agarwal D, Gelman R, Prospero Ponce C, Stevenson W, Christoforidis JB. The Vitreomacular Interface in Diabetic Retinopathy. J Ophthalmol. 2015;2015:392983. doi: 10.1155/2015/392983. Epub 2015 Sep 3. PMID 26425349
- [Background] Duker JS, Kaiser PK, Binder S, de Smet MD, Gaudric A, Reichel E, Sadda SR, Sebag J, Spaide RF, Stalmans P. The International Vitreomacular Traction Study Group classification of vitreomacular adhesion, traction, and macular hole. Ophthalmology. 2013 Dec;120(12):2611-2619. doi: 10.1016/j.ophtha.2013.07.042. Epub 2013 Sep 17. PMID 24053995
- [Background] Yamamoto T, Akabane N, Takeuchi S. Vitrectomy for diabetic macular edema: the role of posterior vitreous detachment and epimacular membrane. Am J Ophthalmol. 2001 Sep;132(3):369-77. doi: 10.1016/s0002-9394(01)01050-9. PMID 11530050
- [Background] Massin P, Audren F, Haouchine B, Erginay A, Bergmann JF, Benosman R, Caulin C, Gaudric A. Intravitreal triamcinolone acetonide for diabetic diffuse macular edema: preliminary results of a prospective controlled trial. Ophthalmology. 2004 Feb;111(2):218-24; discussion 224-5. doi: 10.1016/j.ophtha.2003.05.037. PMID 15019365
- [Background] Dowler JG. Laser management of diabetic retinopathy. J R Soc Med. 2003 Jun;96(6):277-9. doi: 10.1177/014107680309600605. No abstract available. PMID 12782691
- [Background] Khattab AAA, Ahmed MM, Hammed AH. Pars plana vitrectomy for tractional diabetic macular edema with or without internal limiting membrane peeling. Med Hypothesis Discov Innov Ophthalmol. 2022 Dec 3;11(3):110-118. doi: 10.51329/mehdiophthal1454. eCollection 2022 Fall. PMID 37641643
- [Background] Marmor MF, Hood DC, Keating D, Kondo M, Seeliger MW, Miyake Y; International Society for Clinical Electrophysiology of Vision. Guidelines for basic multifocal electroretinography (mfERG). Doc Ophthalmol. 2003 Mar;106(2):105-15. doi: 10.1023/a:1022591317907. No abstract available. PMID 12678274